CLINICAL TRIAL: NCT04652349
Title: A Randomized, Double-Blinded, Multi-center, Phase 3 Study to Evaluate Efficacy and Safety of HGP1910 and HCP1903 in Patients With Primary Hypercholesterolemia
Brief Title: Efficacy and Safety of HGP1910 and HCP1903 in Patients With Primary Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-ROZE-302
Record Dates: First submitted 2020-11-26; First posted 2020-12-03 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Primary Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- HGP1910 (Experimental)
  Interventions: Drug: HGP1910
- HCP1903 (Experimental)
  Interventions: Drug: HCP1903
- HGP1909 (Active Comparator)
  Interventions: Drug: HGP1909
- HGP1911 (Active Comparator)
  Interventions: Drug: HGP1911

INTERVENTIONS:
Drug: HGP1910 — Take it once daily for 8 weeks orally.
  Arms: HGP1910
Drug: HCP1903 — Take it once daily for 8 weeks orally.
  Arms: HCP1903
Drug: HGP1909 — Take it once daily for 8 weeks orally.
  Arms: HGP1909
Drug: HGP1911 — Take it once daily for 8 weeks orally.
  Arms: HGP1911

SUMMARY:
The purpose of this study is to investigate the safety and clinical efficacy of HGP1910 and HCP1903 in patients with primary hypercholesterolemia

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 19 years
* Participants who have voluntarily given written consent to participate in this clinical trial
* Participants with LDL-C ≤ 250mg/dL and TG < 500mg/dL at Visit 1
* Participants with LDL-C ≤ 250mg/dL, TG < 500 mg/dL and satisfied criteria according to cardiovascular risk category at Visit 2 (after at least 4 weeks of TLC)

Exclusion Criteria:

* Patients with active liver disease and severe liver impairment
* Patients with severe renal failure (eGFR < 30 mL/min/1.73 m2 at Visit 1)
* Patients with type I diabetes or uncontrolled type 2 diabetes
* Patients with acute hypertension or uncontrolled hypertension (sitSBP ≥ 180 mmHg or sitDBP ≥ 110 mmHg at Visit 1)
* Patients with symptomatic orthostatic hypotension
* Patients with NYHA class III~IV heart failure, CCSA class III~IV angina, ventricular arrhythmia, severe hemorrhagic or ischemic cerebrovascular diseases, transient ischemic attacks (TIAs), acute coronary syndrome or a history of angioplasty, percutaneous coronary intervention, or coronary artery bypass surgery within six months before Visit 1.
* Patients who were diagnosed with a malignant tumor within five years before Visit.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2020-12-17 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Percentage change(%) from baseline in LDL-C at week 8 | baseline, 8 weeks

SECONDARY OUTCOMES:
Percentage change(%) from baseline in LDL-C at week 4 | baseline, 4 weeks
Percentage change(%) from baseline in LDL-C, TC, HDL-C, non-HDL-C | baseline, 4 weeks, 8 weeks
Percentage change(%) from baseline in Apo A1, Apo B, lipoprotein (a) | baseline, 4 weeks, 8 weeks
Proportion of subjects achieving LDL-C treatment goals by cardiovascular Risk Category | baseline, 4 weeks, 8 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee SA, Kim W, Hong TJ, Ahn Y, Kim MH, Hong SJ, Kim BS, Kim SY, Chae IH, Kim BJ, Rhee MY, Shin JH, Kang TS, Cho JM, Kim JS, Lee CW. Effects of Fixed-dose Combination of Low-intensity Rosuvastatin and Ezetimibe Versus Moderate-intensity Rosuvastatin Monotherapy on Lipid Profiles in Patients With Hypercholesterolemia: A Randomized, Double-blind, Multicenter, Phase III Study. Clin Ther. 2021 Sep;43(9):1573-1589. doi: 10.1016/j.clinthera.2021.07.016. Epub 2021 Aug 21. PMID 34429197